CLINICAL TRIAL: NCT02605408
Title: A Phaco ± LenSx® Procedure Patients Registry in Indian Tertiary Medical Centers
Brief Title: Cataract Surgery in Indian Patients With or Without LenSx® Laser
Status: Withdrawn | Type: Observational
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CTI742-P001
Record Dates: First submitted 2015-11-06; First posted 2015-11-16 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cataract surgery: Phacoemulsification and artificial IOL implantation with and without LenSx® laser system
  Interventions: Device: LenSx® laser system; Procedure: Phacoemulsification

INTERVENTIONS:
Device: LenSx® laser system — Femtosecond laser system used for cornea incision, capsulotomy and lens fragmentation during cataract surgery
Procedure: Phacoemulsification — Removal of the cataractous lens

SUMMARY:
The purpose of this study is to record and analyze the profile and outcome of cataract patients receiving phacoemulsification (phaco) and artificial intraocular lens (IOL) implantation with or without femtosecond laser-assisted cataract surgery (FLACS) in Indian tertiary medical centers.

DETAILED DESCRIPTION:
Legitimate patients will receive Standard of Care (SOC) phacoemulsification treatment for cataract and IOL implantation, with or without using LenSx® technology, with followup for 1 month using SOC postsurgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Agree to undergo phacoemulsification cataract surgery in at least 1 eye;
* Understand and sign an informed consent form;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Refuse to sign the informed consent form or have incomplete medical records;
* Contraindications for phacoemulsification treatment per Investigator discretion or listed in LenSx® Operator's Manual;
* Contraindications for anterior capsulotomy, phacofragmentation of the lens using the FLACS;
* Other protocol-specified exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with cataracts who are receiving phacoemulsification (with or without LenSx® procedure) consecutively during the registry period
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Completion rate of an anterior capsulotomy | Day 0, operative day
Best Corrected Visual Acuity (BCVA) | Up to Day 30 postoperative
Uncorrected Visual Acuity (UCVA) | Up to Day 30 postoperative
Cumulative dissipated energy (CDE) | Day 0, operative day
  Cumulative Dissipated Energy (the amount of ultrasound energy entering the eye during the removal of the cataractous lens) will be reported on the Vision System interface and measured in percent-seconds.
Total phaco + IOL time | Day 0, operative day
Aspiration fluid (ml) | Day 0, operative day
Success rate of IOL insertion | Day 0, operative day
Completion rate of cornea incision | Day 0, operative day
Laser procedure time from suction on to off | Day 0, operative day

CONTACTS AND LOCATIONS:
Overall Officials: Head Medical Affairs, MD, Study Director — Alcon India Pvt. Ltd.